CLINICAL TRIAL: NCT06100731
Title: Evaluating the Impact of Transcranial Direct Current Stimulation on Inhibitory Control in PTSD
Brief Title: tDCS and Inhibitory Control in PTSD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gopalkumar Rakesh (Other)
Responsible Party: Sponsor-Investigator, Gopalkumar Rakesh, Assistant Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 88372
Record Dates: First submitted 2023-10-04; First posted 2023-10-25 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Post Traumatic Stress Disorder
Keywords: noninvasive brain stimulation; inhibitory control; transcranial direct current stimulation
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: Subjects will be randomly assigned to receive Active (real) or Sham (placebo) transcranial direct current stimulation.
Who Masked: Participant, Investigator
Masking Description: Randomization (stratified by PTSD status and medication use) into active or shame tDCS. Double blind software will be used to ensure that the experimenter and the subject remain blind during task administration.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active tDCS (Active Comparator): Current will be ramped in/out for 15 seconds at the beginning and end of a 15-minute period and a constant current will be delivered for the 15-minutes between ramping
  Interventions: Device: tDCS
- Shame tDCS (Sham Comparator): Current will be ramped in/out for 15 seconds at the beginning and end of a 15-minute period during which no stimulation will be delivered.
  Interventions: Device: tDCS

INTERVENTIONS:
Device: tDCS — Subjects will receive 20 minutes of multifocal transcranial direct current stimulation. The anode will be placed over the frontal pole (FC6, 10-10 EEG) and will be surrounded by 5 return electrodes (cathodes). Current will be set at 1.5mA and will be ramped in/ out at the beginning and end of the 15-minutes of stimulation over the course of 15 seconds.
  Other Names: Starstim®; transcranial direct current stimulation; transcranial electrical stimulation

SUMMARY:
Large samples (~2,000/yr) of adult undergraduate students at a large southern university will be pre-screened via the University of Kentucky SONA System (IRB#43626) to identify and recruit adult female participants who report a history of IPV and probable PTSD to participate in a one-day lab study. After completing an IRB-approved informed consent, participants will complete a brief psychiatric diagnostic interview and a battery of questionnaires. They will then complete three blocks of the Stop Signal Task (SST). Participants will be randomized (double-blind, stratified by PTSD diagnosis and psychotropic medication use) to receive 15-min of active or sham multifocal tDCS targeting the rIFG. tDCS will be delivered offline for 11.5-mins after block 1 of the SST and online for 3.5-mins during block 2 of the SST. Sham stimulation will be identical to active tDCS, but electrical current will only be ramped in/out at the beginning and end of the 15-mins. The third block of the SST will be completed after tDCS. Lastly, participants will complete a pictorial trauma-related symptom provocation task. Participants will be compensated with course credit.

DETAILED DESCRIPTION:
Inhibitory control deficits may be a hallmark neuropsychological feature of posttraumatic stress disorder (PTSD). Right inferior frontal gyrus (rIFG) activation is associated with stop signal reaction time (SSRT) - a common measure of inhibitory control - in healthy controls and PTSD patients. PTSD patients exhibit hypoactivation of the rIFG during inhibitory control tasks compared to healthy controls. Moreover, individuals with PTSD may exhibit difficulty modulating rIFG activity in response to increased inhibitory control demands.

The rIFG is also implicated in emotional expression and inhibition. For example, rIFG lesions are associated with difficulty modulating emotional responses and several imaging studies have found that rIFG activity is positively associated with conscious inhibition of negative affect. Among individuals with PTSD, rIFG activity is negatively associated with the severity of PTSD symptoms and the severity of re-experiencing and dissociative symptoms during symptom provocation tasks.

A recent meta-analysis indicates that a single-session of bipolar, anodal (excitatory) neuromodulation of the rIFG with transcranial direct current stimulation (tDCS) can significantly improve SSRT performance (g=0.32). Additionally, multiple studies suggest that anodal tDCS of the rIFG reduce fearful responding to threatening stimuli among psychiatrically healthy participants. One study has examined the effects of tDCS targeting the rIFG on inhibitory control and psychiatric symptoms among a clinical sample that included PTSD patients. Although tDCS did not significantly impact inhibitory control in this study, the use of a mixed psychiatric sample and imprecise tDCS procedures make interpretations difficult. Research has yet to test the effects of tDCS targeting the rIFG on inhibitory control or emotional reactivity in individuals with PTSD.

The proposed study would be the first to explore the effects of multifocal tDCS on inhibitory control and emotional reactivity to trauma cues in a sample of individuals with probable PTSD. This study would contribute to a growing body of evidence showing that tDCS can improve cognitive functioning and influence the expression and inhibition of emotions. Findings may support future research exploring rIFG neuromodulation as an adjunctive treatment for PTSD or a preventative intervention following trauma exposure.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to provide informed consent
2. Ability and willingness to perform procedures
3. Age 18-55
4. Female sex
5. Meet diagnostic criteria for past-month probable IPV-related PTSD.
6. Medication free or stable (≥4 weeks) medication(s)

Exclusion Criteria:

1. Unstable medical, psychiatric, or neurological condition that may necessitate urgent treatment
2. Contraindications for tDCS
3. History of psychosis, mania, major neurological disorder, significant head trauma, or epilepsy.
4. Daily use of psychostimulant medication
5. Daily use of medications that significantly lower seizure threshold
6. Current suicidal intent
7. History of seizures
8. Current pregnancy
9. Moderate severity substance-use disorder

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2023-10-27 (Actual); Primary Completion 2024-12-04 (Actual); Study Completion 2024-12-04 (Actual)

PRIMARY OUTCOMES:
Stop Signal Reaction Time (SSRT) | Day 1
  SSRT is a measure of inhibitory control that is calculated by subtracting the mean stop signal delay on "stop" trials from the mean response time on "go" trials
Skin conductance level (SCL) | Day 1
  SCL will be measured by collecting electrodermal activity (EDA) on the left hand. Mean SCL during trauma related images will be utilized as a measure of emotional reactivity to trauma-related images.
Heart Rate (HR) | Day 1
  HR will be measured using a photophylesmograph on the left hand. Mean HR during trauma related images will be utilized as a measure of emotional reactivity to trauma-related images.

CONTACTS AND LOCATIONS:
Overall Officials: Gopalkumar Rakesh, PhD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: Yes
Upon data de-identification, data will be available upon request after study publication. Upon request, other supporting documents (e.g., study protocol and analytic code) will also be available
Supporting Information: Study Protocol, ICF
Time Frame: May 2025 for 9 years.
Access Criteria: * Must be a doctoral-level researcher.
  * Must request documents from the PI or Co-I of the study.